CLINICAL TRIAL: NCT04752059
Title: Phase II Study of Trastuzumab-Deruxtecan (T-DX; DS-8201a) in HER2-positive Breast Cancer Patients With Newly Diagnosed or Progressing Brain Metastases
Brief Title: Phase II Study of T-DX in HER2-positive Breast Cancer Brain Metastases
Acronym: TUXEDO-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Principal Investigator, Rupert Bartsch, Consultant Medical Oncology, Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TUXEDO-1
Record Dates: First submitted 2021-01-26; First posted 2021-02-12 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Breast Cancer Stage IV
MeSH Terms: conditions — Breast Neoplasms | interventions — trastuzumab deruxtecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- T-DXd 5.4 mg (Experimental): Single arm phase II trial
  Interventions: Drug: Trastuzumab deruxtecan

INTERVENTIONS:
Drug: Trastuzumab deruxtecan — Trastuzumab-deruxtecan 5.4 mg/kg body weight i.v. on day 1 once every three weeks until progression or death
  Other Names: Ds8201a; Enhertu

SUMMARY:
Trastuzumab-Deruxtecan (T-DXd; DS-8201a) in HER2-positive Breast Cancer Patients with newly diagnosed or progressing Brain Metastases

DETAILED DESCRIPTION:
T-DXd will be administered at a dose of 5.4 mg/kg body weight once every three weeks in patients with newly diagnosed or progressive HER2 positive breast cancer brain metastases. Response rate by RANO-BM is defined the primary study endpoint.

ELIGIBILITY:
Inclusion Criteria:

Histologically confirmed breast cancer

* Radiologically documented metastatic disease
* HER2-positive as defined by IHC 3+ and/or HER2/neu gene amplification
* Newly diagnosed brain metastases or brain metastases progressing after prior local therapy
* Measurable disease (RANO-BM criteria)
* No indication for immediate local treatment
* No indication of leptomeningeal disease
* KPS >70%, ECOG <2
* Indication for systemic anti-HER2 treatment
* Prior exposure to trastuzumab and pertuzumab
* Prior exposure to T-DM1 allowed
* Life expectancy of at least 3 months
* Age ≥18 years
* Patient must be able to tolerate therapy, and have adequate cardiac function (defined by baseline left ventricular ejection fraction ≥50%) Adequate bone-marrow, liver and kidney function
* Adequate treatment washout period before enrolment, defined as:
* Major Surgery: ≥4 weeks
* Radiation therapy: ≥4 weeks
* Chemotherapy, small-molecule targeted agents, anticancer hormonal therapy: ≥3 weeks
* Antibody-based treatment: ≥4 weeks
* Patient must be capable of understanding the purpose of the study and have given written informed consent

Exclusion Criteria:

Metastatic breast cancer other than HER2-positve disease

* Use of any investigational agent within 28 days prior to initiation of treatment
* History of malignancy other than squamous cell carcinoma, basal cell carcinoma of the skin or carcinoma in situ of the cervix within the last 3 years including contralateral breast cancer
* Major surgery, other than diagnostic surgery, within the last 4 weeks
* Indication for immediate local therapy as defined by local standard
* Leptomeningeal involvement
* Other anticancer therapy, including cytotoxic, targeted agents, immunotherapy, antibody, retinoid, or anti-cancer hormonal treatment
* Concomitant radiotherapy
* Prior radiotherapy to the thorax other than breast irradiation or irradiation of bone metastases
* A history of uncontrolled seizures, central nervous system disorders or psychiatric disability judged by the investigator to be clinically significant and adversely affecting compliance to study drugs Clinically significant cardiac disease including unstable angina, acute myocardial infarction within six months prior to randomization, congestive heart failure (NYHA III-IV), left ventricular ejection fraction <50%, arrhythmia unless controlled by therapy, with the exception of extra systoles or minor conduction abnormalities, and long QT syndrome (QTc interval >450 ms)
* Subjects who have current active hepatic or biliary disease (with exception of patients with Gilbert's syndrome, asymptomatic gallstones, liver metastases or stable chronic liver disease per investigator assessment) including acute and chronic infections with hepatitis B and C
* Inadequate haematological status at baseline prior to study entry: Dependency on red blood cell and/or platelet transfusions, ANC (absolute neutrophil count (segmented + bands) <1.0 x 109/L; platelets <100 x 109/L
* Inadequate kidney function: serum-creatinine >1.5 times upper normal Limit Hepatic dysfunction: total bilirubin >1.5 times upper normal limit (>3 in patients with liver metastases or known history of Gilbert's disease); ALT, AST >3 times TUXEDO-1_Version 2.0 05.05.2020 Page 8 of 73 upper normal limit (>5 in patients with liver metastases); serum albumin <2.5 g/dL; INR ≥1.5
* Clinically severe pulmonary compromise resulting from intercurrent pulmonary illnesses including, but not limited to, any underlying pulmonary disorder (i.e. pulmonary emboli within three months of the study enrolment, severe asthma, severe COPD, restrictive lung disease, pleural effusion etc.), and any autoimmune, connective tissue or inflammatory disorders with pulmonary involvement (i.e. rheumatoid arthritis, Sjogren's syndrome, sarcoidosis etc.), or prior pneumonectomy.

Subjects with bronchopulmonary disorders who require intermittent use of bronchodilators (such as albuterol) will not be excluded from this study

* Patients with active opportunistic infections
* Known HIV infection
* Concomitant treatment with chloroquine or hydroxychloroquine
* Pregnant or lactating women. Women with childbearing potential must have a negative pregnancy test at screening
* Women with childbearing potential, including women whose last menstrual period was less than one year prior to screening, unable or unwilling to use adequate contraception from study start to one year after the last dose of protocol therapy. Acceptable contraception methods included the application of an intrauterine device, barrier method or total abstinence
* Patients with known hypersensitivity to trastuzumab
* Patients not able to provide written informed consent Patients with known substance abuse or any other medical conditions such as clinically significant cardiac or psychological conditions, that may, in the opinion of the investigator, interfere with the subject's participation in the clinical study or evaluation of the clinical study results
* Patients requiring concomitant use of chronic systemic (IV or oral) corticosteroids at doses higher than 4 mg dexamethasone per day or other immunosuppressive medications except for managing adverse events (inhaled steroids or intra articular steroid injections are permitted in this study)

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-07-28 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Reponse rate of brain metastases to trastuzumab-deruxtecan | From date of randomization until the date of first documented progression or date of death from any cause or treatment discontinuation from any other reason, whichever came first, assessed up to 36 months
  measured according to RANO-BM criteria

SECONDARY OUTCOMES:
Progression-free survival | From date of randomization until the date of first documented progression or date of death from any cause or treatment discontinuation from any other reason, whichever came first, assessed up to 36 months
  Time from inclusion until progression
Overall Survival | From date of randomization until the date of first documented progression or date of death from any cause or treatment discontinuation from any other reason, whichever came first, assessed up to 36 months
  Time from inclusion until death of any cause
Safety of trastuzumab deruxtecan in patients with active brain metastases | From date of randomization until the date of first documented progression or date of death from any cause or treatment discontinuation from any other reason, whichever came first, assessed up to 36 months
  Assessment of treatment-emerging adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Rupert Bartsch, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- AKH Universitaetsklinikum Vienna, Department f. Internal medicine I, oncology, Vienna, Austria

REFERENCES:
- [Result] Bartsch R, Berghoff AS, Furtner J, Marhold M, Bergen ES, Roider-Schur S, Starzer AM, Forstner H, Rottenmanner B, Dieckmann K, Bago-Horvath Z, Haslacher H, Widhalm G, Ilhan-Mutlu A, Minichsdorfer C, Fuereder T, Szekeres T, Oehler L, Gruenberger B, Singer CF, Weltermann A, Puhr R, Preusser M. Trastuzumab deruxtecan in HER2-positive breast cancer with brain metastases: a single-arm, phase 2 trial. Nat Med. 2022 Sep;28(9):1840-1847. doi: 10.1038/s41591-022-01935-8. Epub 2022 Aug 8. PMID 35941372

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-05): https://cdn.clinicaltrials.gov/large-docs/59/NCT04752059/Prot_SAP_000.pdf